CLINICAL TRIAL: NCT02435108
Title: A Pilot Study of Crizotinib in Patients With c-MET Positive Gastric Adenocarcinoma as a Third-line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD, PhD, Division of hematology-oncology, Department of medicine,, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-03-117-003
Record Dates: First submitted 2015-01-15; First posted 2015-05-06 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: c-MET Positive Gastric Cancer
Keywords: MET poisitivity is defined as at least half of tumor cells show weak, moderate or high staining
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- crizotinib arm (Experimental): crizotinib medication
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — crizotinib 250mg bid daily

SUMMARY:
This is a pilot study of crizotinib in patients with c-MET positive gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Advanced gastric adenocarcinoma (including GEJ) that has progressed during or after second line therapy.
4. c-MET positive gastric cancer
5. ECOG PS 0-2
6. At least one measurable disease
7. Proper organ function

Exclusion Criteria:

1. severe co-morbid illness and/or active infections
2. pregnant or lactating women
3. History of documented congestive heart failure; angina pectoris requiring medication; evidence of tranasmural myocardial infarction on ECG; poorly controlled hypertension; clinically significant valvular heart disease; or high risk of uncontrollable arrhythmia
4. active CNS metastases not controllable with radiotherapy or corticosteroids (however, CNS metastases (except for leptomeningeal seeding) are allowed if controlled by gamma knife surgery or surgery or radiotherapy or steroid)
5. known history of hypersensitivity to study drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
progression-free survival | expected average of 24 weeks

SECONDARY OUTCOMES:
overall response rate | up too 100 weeks
overall survival | up too 100 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up too 100 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical center, Seoul, South Korea